CLINICAL TRIAL: NCT05083767
Title: Effect of Whole Body Vibration Training on Glycemic Control in Type II Diabetic Patients: A Randomized Control Trial
Brief Title: Effect of Whole Body Vibration Training on Glycemic Control in Type II Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ameen Medical and Dental Center (Other)
Responsible Party: Principal Investigator, Sobia Hasan, Principal Investigator, Ameen Medical and Dental Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AmeenMDC
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration (Experimental)
  Interventions: Other: Experimental
- Control Group (Placebo Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The study protocol of WBV includes twelve weeks of whole-body vibration training provided to the Type 2 diabetic patients. It was recommended to all participants that they follow their regular diet and medication during the training. Two sets of six 1-minute vibration squats were designed with 20 seconds of rest, 3 times weekly for a duration 12 weeks (total workout time 36 minutes a week), using a vertical vibration machine. The six static positions consisted of (a) a deep squat position (knee angle 900) (b) an elevated squat position (knee angle 1250) (c) an elevated squat position (with elevated heels) (d) a slight knee flexion1 (hand straps with shoulder bending) (e) a slight knee flexion (hand straps with shoulder abduction) and (f) a slight knee flexion 3 (hand straps with elbow flexion). The training load steadily increased from the initial vibration of 30 Hz and the platform amplitude was raised from 2 mm at week 1 to 40 Hz and from 4 mm at week 5 to the completion of training.
  Arms: Whole Body Vibration
Other: Control — The control group was advised to their normal physical activity level, diet, and medication.
  Arms: Control Group

SUMMARY:
Worldwide, the non-communicable diseases are increasing at an alarming rate in which the cardiovascular diseases and Diabetes Mellitus (DM) are predominantly common in lower middle income countries. According to Center of Disease Control and Prevention, Diabetes Mellitus (DM) is the 7th leading cause of mortality in United States that may leads to visual deficits, limb amputations, and organ failure. The prevalence of diabetes in the last few decades has increased along with obesity. According to World Health Organization (WHO) the world wide prevalence of DM has increased up to 422 million people and out of this majority lived in the low-and middle income countries. Almost 1.6 million of death is directly attributed to diabetes. According to International Diabetic Foundation, by the end of 2040, DM will affect up to 642 million of the world population. In Pakistan, WHO reported that 12.9 million patients (10% of the population) have diabetes, 9.4 million patients have diagnosed diabetes, and 3.5 million have not been diagnosed. On the contrary, 38 million people have prediabetes (20.5% women and 15.9% men). Another research has shown that Pakistan is ranked on 7th out of 10 countries with Type II diabetes and will be 4th by 2030. Moreover, about 120,000 people in Pakistan have been reported to die each year as the result of type II diabetes and relative complicated diseases. The keystone of diabetes management includes pharmacological management and changes in the lifestyle that includes physical activity and diet. Regular exercises not only improve the cardiovascular fitness but also help in improving the regulation of blood glucose there by enhance insulin signaling, improved vascular function and blood lipids, as well as reduced low-grade inflammation, and weight loss. Researchers suggested that physical activity can boost insulin sensitivity for patients with type II diabetes and help to reduce high blood glucose levels. During exercise, the intake of oxygen can increase up to 20 times and is greatly increased in working muscles. However, receptivity to perform exercises among general population is poor; mainly due to substantial commitment of time associated in performing these exercises. As a passive interference, therefore, Whole-body vibration (WBV) was introduced. Vibration training elevates, energy utilization and increases the blood flow of periphery. Hence the current study was focused on examining the effects of WBV on HbA1c and Fasting Blood Sugar (FBS) in type II diabetic patients.

DETAILED DESCRIPTION:
A double-blinded randomized controlled trial was conducted among type-II diabetic patients; aged 40-70 years recruited between April 2019 to May 2020 using simple random sampling technique's envelope method from a primary care center of Karachi. All the participants were initially screened by two certified diabetes educators and certified health fitness programmers. Participants were given informed consent prior to intervention, their voluntary participation and understanding of the protocol was ensured prior to the commencement of protocol.

Participants who met the inclusion criteria were assigned by computer-generated number into two groups A and B (n=15) in each group. Group A was provided with Whole Body Vibration (WBV) for twelve weeks whereas Group B (control group) was instructed to continue their medications and dietary plan. The outcome measure of the study was FBS and HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Age between 40-70 years

Exclusion Criteria:

* Diagnosed neurological and cardiovascular condition
* Untreated orthostatic hypotension
* unwilling to participate

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
HbA1c | Baseline
HbA1c | 12 weeks
Fasting Blood Sugar | Baseline
Fasting Blood Sugar | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sobia Hasan, MS, Principal Investigator — Ameen Medical and Dental Center
Locations (1):
- Ameen Medical and Dental Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No